CLINICAL TRIAL: NCT03033537
Title: Intracavernosal Injection of Papaverine/Verapamil Versus Papaverine/Phentolamine in Erectile Dysfunction: A Pilot Study
Brief Title: Intracavernosal Injection of Papaverine/Verapamil Versus Papaverine/Phentolamine in Erectile Dysfunction
Status: Completed | Type: Observational
Sponsor: Adam International Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Raef Sadek, Dr., Adam International Hospital
Other Study IDs: 2016
Record Dates: First submitted 2017-01-20; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Verapamil; Calcium Channel Blockers

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Verapamil: Intracavernosal injection of Verapamil
  Interventions: Drug: Verapamil
- Phentolamine: Intracavernosal injection of Phentolamine to treat erectile dysfunction for a period of 2 wweks
  Interventions: Drug: Verapamil

INTERVENTIONS:
Drug: Verapamil — Local treatment of erectile dysfunction
  Other Names: Calcium Channel Blocker

SUMMARY:
Introduction: Erectile dysfunction is a common condition with a significant effect on quality of life. Verapamil is calcium channel blocker of the phenyl alkylamine class which relaxes the tone of the smooth muscles lining blood vessels, leading to their dilatation.

DETAILED DESCRIPTION:
Objective: Evaluating the effect of intracavernosal injection of (Papaverine + Verapamil) and comparing it with (Papaverine + Phentolamine) in patients with erectile dysfunction.

Patients and methods: Each one of the 20 erectile dysfunction patients was subjected to intracavernosal injection with (30mg Papaverine + 1mg Phentolamine), where penile duplex & clinical evaluation was carried out followed by a wash out interval of 2 weeks after which each patient was subjected to the exact previous procedures using (30 mg Papaverine + 5 mg Verapamil).

Keywords: Erectile dysfunction - Intracavernosal injection - Penile duplex - Phentolamine - Verapamil.

ELIGIBILITY:
Inclusion Criteria:

* Married male patients suffering from erectile dysfunction and scheduled for intracavernosal injection.

Exclusion Criteria:

* Responders to PDE5-inhibitors; congenital or acquired penile anomalies; uncontrolled medical conditions or known hypersensitivity to verapamil; Peyronie's disease and any known bleeding or coagulation disorders.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Males complaining of erectile dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-20 (Actual)

PRIMARY OUTCOMES:
IIEF5 | 6 months
  Questionnaire

IPD SHARING:
Plan to Share IPD: No